CLINICAL TRIAL: NCT06996626
Title: Real-time Evaluation of an Outlier-based Alerting System
Brief Title: Real-time NOMA Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David T Huang (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor-Investigator, David T Huang, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25020040; 5R01EB032752-10 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Step wedge RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Unrevealed Alerts (Active Comparator)
  Interventions: Device: Unrevealed Alerts
- Revealed Alerts (Experimental)
  Interventions: Device: Revealed Alerts

INTERVENTIONS:
Device: Revealed Alerts — Bedside reveal of alerts generated by the alerting system
  Arms: Revealed Alerts
Device: Unrevealed Alerts — Alerts will be generated but not revealed.
  Arms: Unrevealed Alerts

SUMMARY:
Alerts related to outlier clinician behavior are generated in real-time by an intelligent system continuously scraping EHR (electronic health record) data. These alerts are passed to the bedside and their potential impact on bedside clinical behavior is evaluated.

DETAILED DESCRIPTION:
A clinician-informed AI model will generate outlier alerts from real-time review of the EHR (electronic health record) of UPMC Presbyterian/Montefiore ICU patients. These alerts will first be reviewed by an ICU clinician, along with the patients' EHR, for clinical relevance. For those alerts deemed potentially relevant, the ICU clinician will contact the treating ICU clinician (eg, an ICU pharmacist, physician, advanced practice provider) and discuss the alert. The treating ICU clinician will take whatever action, including no action, they deem best.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the Presbyterian and Montefiore ICUs

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Actions Following Revealed vs. Non-Revealed Alerts | From time of ICU admission until ICU discharge
  The primary outcome compares the proportion of alerts that lead to documented clinical actions when revealed to treating ICU clinicians versus when not revealed. Alerts are generated by a decision support system and reviewed daily by ICU study clinicians. On average, 30 alerts are reviewed per ICU per day, with approximately 5 alerts revealed to the treating clinicians. The analysis uses a stepped wedge design with ICU beds as the unit of analysis, where each ICU acts as its own control. The outcome will assess whether revealing alerts increases the rate of appropriate clinical actions taken, as compared to when alerts are withheld.

SECONDARY OUTCOMES:
Rate of Any Clinically Responsive Action Following Alerts | Up to 90 days after ICU admission
  For each alert, a range of clinical actions may be deemed "responsive," including but not limited to the specific recommended action. This outcome assesses the differential rate of any clinically appropriate response (whether or not it matches the recommended action) between alerts that are revealed versus not revealed to treating ICU clinicians.
True Positive Alert Rate (TPAR) by Study Group and Alert Type | Up to 90 days after ICU admission
  This outcome evaluates the overall and alert-specific True Positive Alert Rate (TPAR), defined as the proportion of alerts that are associated with a clinically appropriate action. TPARs will be calculated separately for the intervention group (alerts revealed), the control group (alerts not revealed), and the combined population. Comparisons will assess whether revealing alerts is associated with a higher TPAR across alert categories.
Rate of Non-Responsive Actions Following Alerts | Up to 90 days after ICU admission
  This outcome assesses the difference in the rate of clinical actions that are not considered responsive to the alert (i.e., actions taken that do not address the alert's content or recommended intervention) between the intervention group (alerts revealed) and the control group (alerts not revealed). This helps evaluate potential unintended or off-target responses to alerting.
Overall Alert Rate | Through study completion, an average of 2 years
  Total number of alerts generated per ICU per day.
Alert Rate per Alerting Model | Daily, up to 90 days
  Number of alerts generated per model type per ICU per day.
Delay Between Alert Generation and First Responsive Action | Measured continuously through study completion, an average of 2 years
  Median time from alert generation to the first documented responsive clinical action.
ICU Length of Stay | Up to 90 days after ICU admission
  Total number of days each participant spends in the ICU during the index hospitalization.
Hospital Length of Stay | up to 90 days after hospital admission
  Total number of days each participant spends in the hospital during the index hospitalization.
In-Hospital Mortality | Up to 90 days after hospital admission
  Proportion of participants who die during the index hospital stay.
Time Trend of True Positive Alert Rate (TPAR) | Through study completion, an average of 2 years
  Evaluate changes in the True Positive Alert Rate (TPAR) over time during the study period to assess model performance stability and potential temporal variation in responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Montefiore, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The investigators do not currently have a data sharing plan for sharing with future investigators. If the investigators decide to share data in the future with investigators conducting similar research both inside and outside of the University of Pittsburgh, the investigators will contact the Office of Sponsored Programs before sharing de-identified research data to determine whether an agreement needs to be executed.